CLINICAL TRIAL: NCT05337306
Title: Increasing Health Equity Through In-The-Moment Reading Assistance for Adults With Diabetes Served at Community Health Centers
Brief Title: Improving Diabetic Patient Health Through Assistive-Reading Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GogyUp Inc (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R43NR020340 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-04-20 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2; Health Knowledge, Attitudes, Practice; Literacy
Keywords: adherence; adult; aftercare; chronic disease; diabetes mellitus; educational materials; health education; Limited English Proficiency; patient education; literacy; health literacy; assistive technology; health disparity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior; Literacy; Chronic Disease; Diabetes Mellitus; Health Education

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GogyUp (Experimental): Participants in the GogyUp arm will have the GogyUp Reader app preloaded on a cellular-enabled tablet with the same patient education documents as the Control arm. Patients will be able to use on-demand / in-the-moment assistive-reading technologies to understand any word or phrase:
  * Speech-to-Text
  * Word-by-Word Translation
  * Alternative Formatting
  * Simplified and Contextualized Definitions
  * No-Fail Comprehension Questions
  * Personalized Training in Phonemic Awareness
  Interventions: Other: GogyUp Reader
- Control (No Intervention): Participants in the Standard Care arm will receive the standard after-visit patient education documents the clinics current provide for type 2 diabetes education and self-management.

INTERVENTIONS:
Other: GogyUp Reader — Participants will have unlimited access to the assistive-reading technologies available in the GogyUp Reader app for help understanding post-visit educational documents on type 2 diabetes mellitus disease management.
  Arms: GogyUp

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) affects over 30 million Americans and requires patients to competently manage their conditions at home. However, the majority of diabetes self-management education (DSME) and aftercare print materials remain overly complicated, with excessively high reading difficulty and fall short in supporting functional readiness for self- management at home, especially for the 18% of U.S. adults unable to read beyond a second-grade level. This project will determine the feasibility of implementing assistive reading technology, designed for patients with limited print or English proficiency, that will immediately expand patient capacity to understand DSME materials, increase T2DM self- management adherence and eventually reduce, at a scale, disparate outcomes in a chronic disease. It will use a small pilot trial design of the GogyUp Reader app to use with print materials versus print materials with no app support and test effects of GogyUp on three-month follow-up measures of health literacy (primary outcome) using the Health Literacy Questionnaire subscales 9 (Understanding health information well enough to know what to do") and 2 ("Having sufficient information to manage my health"); and on three-month follow-up self-reported diabetes management (secondary outcome) using the Perceived Diabetes Self-Management Scale (PDSMS).

DETAILED DESCRIPTION:
Diabetes self-management requires knowledgeable communication and capacity for self-management. People with type 2 diabetes mellitus (T2DM) must learn from health care providers about the condition to build knowledge on how to manage the disease and competently carry out self-management. T2DM self-management is extensive: estimates of time spent on recommended self-management activities can exceed 10 hours per week, equivalent to part-time employment. Effective T2DM-related self-management requires patients to read, understand, and execute care plans. In short, T2DM comes with a demanding workload that assumes patients have enough capacity to read and follow complex instructions to successfully manage their disease.

Barriers to building understanding and competence for self-management both reflect and contribute significantly to inequality. Existing social systems in the United States have provided inequitable educational achievement, including literacy in general and health literacy in particular. The result is that the U.S. has widespread and entrenched adult illiteracy. 18% of U.S. adults (roughly 44 million) are unable to decipher unfamiliar words or identify information in short texts. In practical terms, a large segment of the U.S. population is without the skills to read medicine or nutrition labels, follow written aftercare instructions, etc. This deficit is reflected in the T2DM patient population. Large percentages (e.g., 35-55%) of individuals with T2DM have reading levels at 6th grade or below, with lower literacy significantly associated with several demographic variables (e.g., lower socioeconomic status), indicating inequitable distribution. Moreover, lower functional English and health literacy, and poorer diabetes knowledge, are associated with poorer glycemic control.

However, work on facilitating the entry of adults with limited literacy and English proficiency into the workforce demonstrates that these challenges can be successfully addressed through an integrated adult literacy approach. This approach of "integrated adult literacy" combines the delivery and understanding of concepts and information with in-the-moment assistive-reading technology and contextualized literacy instruction regardless of whether an adult employee is correctly perceived to be at risk for missing critical information.

Health care supports for capacity in self-management lack appreciation for integrated adult literacy and have limited effectiveness. Health literacy is not only an individual issue, but also reflects if systems and materials are calibrated to individual capacity. Yet health care does not typically operate in recognition of this fact. Written patient materials for post-visit care are consistently complex, often far exceeding the intended consuming audience's reading level. Meanwhile, practices such as "Teach Back" and including interpreters in clinic visits have short-term benefits for patient understanding and ability to carry out self-management; as these effects diminish over time, mastery of key information becomes elusive. The inadequacy of these measures is compounded by stigma that can accompany low literacy or limited English proficiency. Even patients who have developed literacy skills may be embarrassed about a lack of understanding. Stigma, embarrassment, or simply the stress of a clinical appointment can prevent patients from asking clarifying or follow-up questions, a process integral to establishing content mastery.

Existing systems are inadequate to bridging gaps in patients' needs and readiness to manage diabetes. Achieving universal literacy in the U.S. adult population historically has been a major challenge; systems in place lack sufficient system capacity and scale to address it. For example, only a fraction of U.S. adults in need of reading instruction have access to it. Literature indicates a growing recognition by health educators of the potential for engaging with and implementing techniques from adult basic education, including integrated adult literacy. However, significant factors would still limit the impact which implementing such measures could have for patients with limited literacy or English proficiency. Foremost would be the significant issue of scale needed for impact and improvement.

A paradigm shift is needed, from clinic-by-clinic intervention to highly scalable, low cost in-the-moment support using assistive technology (AT) but little is known, particularly from an integrated adult literacy perspective. As noted, existing systems are inadequate to increase integrated adult literacy generally, and clinical interventions require patients to retain knowledge as they use complex, written instructions and education materials in self-management away from the clinic. Because changes to these have historically remained out of reach, the investigators propose shifting the paradigm away from focusing on providers' capacity to communicate and educate, and toward supporting patients' capacity to access, comprehend and internalize health education through AT, expanding their capacity for self-management in the moment, on an as-needed basis. AT commonly refers to any equipment, software, etc. that is used to maintain or improve the functional capabilities of individuals with disabilities, often with features and functions that can be adjusted to an individual's specific requirements. Notably, existing electronic health (eHealth) and mobile health (mHealth) support technologies with text-heavy interfaces have not incorporated reading AT and are frequently limited to single-use applications with poor readability, and/or usability issues, negating their benefit for integrated adult literacy for diabetes self-care.

Substantial evidence describes how AT equalizes information access across education levels. When combined with the near-ubiquity of mobile devices and telecommunications networks, AT - and specifically assistive reading technology - holds the potential for universal, integrated adult literacy supports that could substantially impact diabetes self-management education. Sidewalk cutouts offer a useful analogy for whole-population benefit. While cutouts expand mobility to those using walkers and wheelchairs, they also provide unintended benefits to any child riding a bicycle or parent pushing a stroller. Similarly, benefits from reading AT could extend beyond the intended population (e.g., adults with limited functional literacy or English proficiency) to those with diminished eyesight and even fully literate adults simply struggling with difficult materials.

The current study will use a small pilot trial design of the GogyUp reader app for use with print materials versus no support for reading capacity among adults with diabetes.

Primary Endpoint: three-month (follow-up) scores on two subscales of the Health Literacy Questionnaire: Subscale 9: Understanding health information well enough to know what to do ("Understanding health information"); Subscale 2: Having sufficient information to manage my health ("Having sufficient information").

Secondary Endpoint: three-month (follow-up) score on the Perceived Diabetes Self-Management Scale (PDSMS).

Analysis: We will compare the mean outcomes at follow-up between the treatment arms using analysis of covariance (ANCOVA), which compares follow-up outcome values between study arms while controlling for the baseline levels to gain power to detect an effect. The primary analysis will be an intent-to-treat (ITT); for non-monotonic missing (e.g., missing a baseline value), we will use multiple imputation with pattern mixture model adjustments in sensitivity analyses allowing for plausible differences among the missing-the justification for this is that pattern mixture models allow for a Missing Not At Random assumption, which is plausible in this case because we will not have measures for all likely variables associated with missingness. Pattern mixture models allow for us to set plausible values for missingness at both high or low levels to obtain a range of outcome estimates allowing for plausible missing data scenarios. For any monotonic missing- i.e., attrition (withdrawal or other lost to follow-up), we will use last observation carried forward but will also conduct sensitivity analyses using pattern mixture models under plausible assumptions of missing data patterns. We will present results using adjusted (least-squares) means with standard errors, p-values, and 95% confidence intervals. Baseline levels of endpoint outcomes will be included as a covariate to gain power to detect an effect, a standard use of ANCOVA.

The maximum sample size is up to 200 individuals, with expectation of potential non-contact by patients after a recruitment mailing, screening failures and refusal bringing likely sample size down to approximately 120-160. The target population are individuals aged 18-85 diagnosed with type 2 diabetes mellitus seen at clinics serving large proportions of low-income patients (e.g., safety net clinics). We will attempt to sample up to 200 individuals from the MHealth Fairview health system in the seven-county Twin Cities Metropolitan area.

Study activities will not take place in any clinical sites; participants will be identified based on having been seen for a clinic visit to a primary care clinic within the partnering health system and will receive a mailing from the health system providing contact information for the researchers; patients will themselves contact the research team if they choose. The study will not include sites outside of the United States.

Contribution: Understanding use and potential benefit of in-the-moment reading support for adult patients in understanding diabetes self-management written materials. The potential benefit of reading AT, readily embedded in adult patients' lives, that expands their capacity to use written materials at scale, at low cost, and particularly from an integrated adult literacy standpoint, has not been previously studied.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Males and females; Aged 18-85 years
3. Documented diagnosis of type II diabetes mellitus
4. Has had a visit to a clinic in the past year (April 2020-February 2021); can include a telehealth visit
5. Receives patient education materials and can consent in English

Exclusion Criteria:

1. Currently enrolled in another treatment or intervention study (at pre-screen)
2. Pregnancy (because pregnancy becomes the primary condition of interest)
3. Note: Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone, internet access) will not be a criterion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ned Zimmerman-Bence, Principal Investigator — GogyUp Inc
Locations (1):
- MHealth Fairview system, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Shippee (having led analyses) will submit summary results to ClinicalTrials.gov following timeline completion of the analyses concurrent with manuscript results preparation, which should be within two to three months post follow-up for final participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study data will be available once final report has been accepted by the National Institute for Nursing Research (the funding agency). Analytic date will remain available through the University of Minnesota's Clinical Data Repository managed by the University of Minnesota's Clinical and Translational Sciences Institute.
Access Criteria: Criteria include employees of federal agencies or institutions of higher learning.

REFERENCES:
- See also: Reference List for Improving Diabetic Patient Health Through Assistive-Reading Technology — https://docs.google.com/document/d/1VummtaTzQ15PlLgNmHM8LCfyp86OSW1NKbDz1xkL3-c/edit?usp=sharing

RESULTS

PARTICIPANT FLOW:
Groups:
- GogyUp: Participants in the GogyUp arm will have the GogyUp Reader app preloaded on a cellular-enabled tablet with the same patient education documents as the Control arm. Patients will be able to use on-demand / in-the-moment assistive-reading technologies to understand any word or phrase:
  * Speech-to-Text
  * Word-by-Word Translation
  * Alternative Formatting
  * Simplified and Contextualized Definitions
  * No-Fail Comprehension Questions
  * Personalized Training in Phonemic Awareness
  GogyUp Reader: Participants will have unlimited access to the assistive-reading technologies available in the GogyUp Reader app for help understanding post-visit educational documents on type 2 diabetes mellitus disease management.
Period: Overall Study
Arm/Group | GogyUp | Control
Started | 101 | 92
Completed | 73 | 70
Not Completed | 28 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GogyUp | Control | Total
Number analyzed (Participants) | 101 | 92 | 193
Age, Categorical [Count of Participants; unit: Participants] — Population: For age: 30 GogyUp participants and 24 Control participants were missing baseline age. Age was not used as a covariate.
  Participants
    number analyzed (Participants) | 71 | 68 | 139
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 32 | 35 | 67
    >=65 years | 39 | 33 | 72
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: For gender, 15 GogyUp and 10 Control participants were missing baseline gender. Gender was not used as a covariate.
  Participants
    Sex not analyzed: number analyzed (Participants) | 86 | 82 | 168
    Sex not analyzed: Female | 49 | 40 | 89
    Sex not analyzed: Male | 36 | 42 | 78
    Sex not analyzed: Prefer not to answer | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Health Literacy Questionnaire subscale 9 [Mean (Standard Deviation); unit: units on a scale] | 4.086 (.395178) | 4.03297 (.43743) | 4.0607 (.415588)
Health Literacy Questionnaire subscale 2 [Mean (Standard Deviation); unit: units on a scale] | 2.8825 (.492949) | 2.777 (.5470) | 2.8324607 (.520697)
Perceived Diabetes Self-Management Scale [Mean (Standard Deviation); unit: units on a scale] — Population: PDSMS measures were missed at baseline for some early participants: 35 GogyUp and 31 Control participants were missing this measure at baseline.
  units on a scale
    number analyzed (Participants) | 66 | 61 | 127
    (all) | 28.136 (5.8936) | 27.295 (6.3727) | 27.73228 (6.118)

OUTCOME MEASURES:

1. Primary Outcome: Health Literacy Questionnaire Subscale 9: Understanding Health Information Well Enough to Know What to do
Description: The first primary outcome is three-month (follow up) value of the Health Literacy Questionnaire (HLQ) subscale 9: Understanding health information well enough to know what to do
  The "Understanding health information" subscale is a multi-item, validated subscale of the HLQ and a continuous variable. It is a 5-item subscale, with items scored 1-5 (with higher scores being better) and then mean-aggregated.
  This study's main objective is to study the effect of GogyUp on health literacy (the ability to use and understand written health information) as a proximal effect of support. The Understanding health information subscale is the most direct measure; three-month follow up reflects (a) brief follow-up in a pilot trial; and (b) this outcome is very proximal to the intervention.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GogyUp | Control
Number analyzed (Participants) | 101 | 92
units on a scale | 4.2079 (.4621) | 4.31739 (.4439)
Statistical Analysis 1: Comparison: GogyUp vs Control; Last Observation Carried Forward (LOCF) for those lost to follow up; null hypothesis group 1 follow-up outcome = group 2 follow-up outcome; Test type: Superiority — ANCOVA controlling for study arm and baseline; p = .049, ANCOVA — a priori threshold .05; no adjustment for multiple comparisons; covariates include arm and baseline level of outcome

2. Primary Outcome: Health Literacy Questionnaire Subscale 2: Having Sufficient Information to Manage my Health
Description: The other primary outcome measurement is the three-month (follow up) value of the validated Health Literacy Questionnaire Subscale 2: having sufficient information to manage my health.
  The "Having sufficient information" subscale is a multi-item, validated subscale of the HLQ and a continuous variable. It is a 4-item subscale, with items scored 1-4 (with higher scores being better) and then mean-aggregated.
  This study's main objective is to study the effect of GogyUp on health literacy (def: the ability to use and understand written health information) as a most proximal effect of in-the-moment support. As such, the Having sufficient information subscale is an additional direct measure; the three-month time frame reflects (a) a brief follow-up as part of a pilot trial; and (b) is reasonable because of the use of this proximal (to the intervention) outcome based on putative mechanisms.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GogyUp | Control
Number analyzed (Participants) | 101 | 92
units on a scale | 3.03465 (.4835) | 3.16304 (.5351)
Statistical Analysis 1: Comparison: GogyUp vs Control; LOCF for lost to follow-up; Test type: Superiority; p = .040, ANCOVA — a priori threshold .05; no adjustment for multiple comparisons; Covariates include trial arm and baseline level of outcome

3. Secondary Outcome: Perceived Diabetes Self-Management Scale Score
Description: The secondary outcome measure is the three month (follow-up) score on the Perceived Diabetes Self-Management Scale (PDSMS)
  PDSMS is a validated measure (continuous variable). It has eight items ranged 1-5 and summed (range 8-40), with higher scores being better.
  This study's objective is to study the effect of GogyUp on health literacy (the ability to use and understand written health information) as a proximal effect of in-the-moment support. However, any benefit is expected to be via translation of improved health literacy into improved diabetes self-management. As such, this secondary outcome is less proximal but still relevant. The three-month time frame reflects brief follow-up as part of a pilot trial but benefit may not accrue within the short timeframe, meaning this measure may be most useful for obtaining effect size estimates to inform sample size calculations for future studies.
Time Frame: 3 months
Population: Some baseline PDSMS scores were not collected at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GogyUp | Control
Number analyzed (Participants) | 88 | 84
units on a scale | 24.3409 (3.12898) | 24.8452 (3.6553)
Statistical Analysis 1: Comparison: GogyUp vs Control; LOCF for dropout/lost to follow up; Test type: Superiority; p = .220, ANCOVA; covariates include trial arm and baseline level of outcome

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | GogyUp | Control
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/92
Other Adverse Events (participants affected / at risk) | 0/101 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT05337306/Prot_SAP_ICF_000.pdf